CLINICAL TRIAL: NCT03649971
Title: A Phase 1b, Multicenter, Randomized, Blinded, Placebo-controlled Study to Evaluate the Efficacy of Guselkumab in Subjects With Familial Adenomatous Polyposis
Brief Title: A Study of Guselkumab in Participants With Familial Adenomatous Polyposis
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Janssen Research & Development, LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CR108515; CNTO1959COR1001 (Other: Janssen Research & Development, LLC); 2019-001980-57 (EudraCT Number)
Record Dates: First submitted 2018-08-27; First posted 2018-08-28 (Actual); Last update posted 2025-02-03 (Actual); Status verified 2025-01

CONDITIONS: Adenomatous Polyposis Coli
MeSH Terms: conditions — Adenomatous Polyposis Coli | interventions — guselkumab

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Guselkumab Dose 1 (Experimental): Participants will receive guselkumab Dose 1 subcutaneous (SC), 6 doses every 4 weeks from Week 0 to Week 20. Participants who respond to guselkumab may continue treatment at the same dose level through Week 48.
  Interventions: Drug: Guselkumab
- Guselkumab Dose 2 (Experimental): Participants will receive guselkumab Dose 2 SC, 6 doses every 4 weeks from Week 0 to Week 20. Participants who respond to guselkumab may continue treatment at the same dose level through Week 48.
  Interventions: Drug: Guselkumab
- Placebo (Placebo Comparator): Participants will receive placebo SC, 6 doses every 4 weeks from Week 0 to Week 20.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Guselkumab — Guselkumab SC will be administered every 4 weeks.
  Other Names: Tremfya
  Arms: Guselkumab Dose 1; Guselkumab Dose 2
Drug: Placebo — Placebo SC will be administered every 4 weeks.
  Arms: Placebo

SUMMARY:
The purpose of this study is to determine the effect of treatment with guselkumab in participants with familial adenomatous polyposis (FAP) on rectal/pouch polyp burden.

DETAILED DESCRIPTION:
Familial adenomatous polyposis (FAP) is the most common polyposis syndrome. It is autosomal dominant inherited disorder characterized by early onset of hundreds to thousands of adenomatous polyps throughout colon. If left untreated, this syndrome may develop colorectal cancer (CRC). Polyps from individuals with FAP display inflammatory features associated with activation of interleukin (IL) 23/IL 17/JAK/STAT3 pathway. This inflammation is thought to contribute to further mutagenesis, culminating in tumor development. Specifically, IL-23 is linked to tumor growth and progression in CRC. Guselkumab is a human immunoglobulin monoclonal antibody directed against p19 subunit of IL-23, specifically targets IL-23 and inhibits its interaction with IL-23 receptor, inhibiting IL 23 specific intracellular signaling and subsequent cell activation and cytokine production, which result in less inflammation and reduce tumor development. The clinical hypothesis of this study is that treatment with guselkumab will reduce rectal/pouch polyp burden compared with baseline in active arms compared with placebo. The study is designed to determine if guselkumab has clinical activity in colorectum and duodenum, by reducing number of polyps over a period of 24 weeks. Participants will be randomized to 1 of 3 treatment arms (Guselkumab 100 mg [milligram] SC [subcutaneous], Guselkumab 300 mg SC, and placebo SC). Efficacy evaluations include rectal/pouch polyp burden assessment, biomarker analysis include discrete IL-23 signaling effector proteins (IL-23R, pSTAT3, Il-17A) and safety evaluations will include monitoring of adverse events, laboratory tests, vital sign measurements, and physical examination. Safety will be monitored throughout study (up to Week 60).

ELIGIBILITY:
Inclusion Criteria:

* Phenotypic familial adenomatous polyposis (FAP) with disease involvement of the colorectum by either genetic or clinical diagnosis: Adenomatous polyposis coli (APC) germline mutation with or without family history, or with greater than (>)100 adenomas in large intestine and a family history of FAP, attenuated FAP is allowed. FAP phenotype post colectomy for polyposis with a family history of FAP may be allowed
* Post-colectomy or subtotal colectomy
* Polyps with a sum of diameters greater than or equal to (>=)10 millimeter (mm) in the rectum or pouch on biopsy at screening
* A woman of childbearing potential must agree not to get pregnant during the study and at least 12 weeks after the last dose of study administration
* A woman must agree not to breast feed or donate eggs (ova, oocytes) during the study and for a period of 12 weeks after the last administration of study drug

Exclusion Criteria:

* Prior use of any biologic therapy targeting interleukin (IL)-12/23, IL-17, or IL-23 receptor
* Use of non-steroidal anti-inflammatory drugs other than aspirin during the study. The use 100 milligram (mg) of aspirin a day or 700 mg of aspirin per week is allowed
* Treatment with other FAP-directed drug therapy (including NSAID [Nonsteroidal anti-inflammatory drug] drugs), unless completes a 4-week washout period prior to randomization
* High grade dysplasia or cancer on biopsy at screening in GI tract (including stomach, duodenum, and colon/rectum/pouch)
* Duodenal, colorectal, or pouch polyp: >2 centimeter (cm) unless excised at the screening evaluation; and 1 to 2 cm with evidence of high-grade dysplasia upon biopsy unless excised

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 77 (Actual)
Dates: Start 2018-11-19 (Actual); Primary Completion 2021-09-13 (Actual); Study Completion 2022-03-23 (Actual)

PRIMARY OUTCOMES:
Percentage Change from Baseline in Rectal/pouch Polyp Burden at Week 24 | Baseline, Week 24
  Percentage change from baseline in rectal/pouch polyp burden (sum of the polyp diameters) at Week 24 will be determined through endoscopy.

SECONDARY OUTCOMES:
Percentage Change from Baseline in Number of Colorectal Polyps | Baseline, Weeks 24 and 52
  Percentage change from baseline in number of colorectal polyps will be determined.
Percentage Change from Baseline in Number of J-pouch Polyps | Baseline, Weeks 24 and 52
  Percentage change from baseline in number of J-pouch polyps will be determined.
Percentage Change from Baseline in J-pouch Polyp Burden | Baseline, Weeks 24 and 52
  Percentage change from baseline in J-pouch polyp burden (sum of polyp diameters) will be determined.
Percentage Change from Baseline in Number of Duodenal Polyps | Baseline, Weeks 24 and 52
  Percentage change from baseline in number of duodenal polyps will be determined.
Percentage Change from Baseline in Duodenal Polyp Burden | Baseline, Weeks 24 and 52
  Percentage change from baseline in duodenal polyp burden (sum of polyp diameters) will be determined.
Change in International Society for Gastrointestinal Hereditary Tumors (InSiGHT) Stage | Baseline, Weeks 24 and 52
  Change in InSiGHT stage will be determined. Various stages of InSiGHT staging system are defined as: Stage 0: 0-10 polyps, all less than (<)5 millimeter (mm); Stage 1: 10-25 polyps, most < 5 mm, none greater than (>) 1 centimeter (cm); Stage 2: 10-25 polyps, any > 1 cm, amenable to complete removal; Stage 3: > 25 polyps amenable to complete removal, or any incompletely removed sessile polyp, or any evidence of High-Grade Dysplasia (HGD), even if completely excised; and Stage 4: > 25 polyps amenable to complete removal, or any incompletely excised sessile polyp showing HGD, any invasive cancer).
Change in Spigelman Stage Score | Baseline, Weeks 24 and 52
  Change in Spigelman stage score will be determined. Spigelman classification system measures risk of developing duodenal cancer in familial adenomatous polyposis (FAP). It has been classified in following stages- Stage 0 (0 points); Stage 1 (1-4 points); Stage 2 (5-6 points); Stage 3 (7-8 points); and Stage 4 (9-12 points). The total score ranges from 0 to 12. Points are accumulated for polyps' number, size, histology and severity of dysplasia. Stage 1 indicates mild disease, whereas stage 3-4 indicates severe duodenal polyposis.
Trough Concentration of Guselkumab | Weeks 0, 4, 8, 12, 16, 20, 24, 32, 40, and 48
  Serum samples will be analyzed to determine trough concentrations of guselkumab using a validated specific, and sensitive method.
Number of Participants with Anti-guselkumab Antibodies | Weeks 0, 4, 8, 12, 16, 20, 24, 32, 40, and 48
  Number of participants with Anti-guselkumab antibodies will be determined.
Anti-guselkumab Antibodies Serum Titers | Weeks 0, 4, 8, 12, 16, 20, 24, 32, 40, and 48
  Serum samples will be screened for antibodies binding to guselkumab and the titer of confirmed positive samples will be reported.
Number of Participants with Adverse Events as a Measure of Safety | From Screening up to 60 Weeks
  An adverse event is any untoward medical event that occurs in a participant administered an investigational product, and it does not necessarily indicate only events with clear causal relationship with the relevant investigational product.
Number of Participants with Vital Sign Abnormalities as a Measure of Safety and Tolerability | From Screening up to 52 Weeks
  Number of participants with vital sign abnormalities will be reported. Vital signs includes temperature, pulse/heart rate, respiratory rate and blood pressure.
Number of Participants with Clinical Laboratory Abnormalities as a Measure of Safety and Tolerability | From Screening up to 52 Weeks
  Number of participants with clinical laboratory abnormalities will be reported. Blood samples for serum chemistry and hematology will be collected at predefined time points for clinical laboratory testing.
Relative Changes to Baseline in Levels of Interleukin (IL)-23 Effector Proteins in Biopsy Tissue | Baseline, Weeks 12, 24, and 52
  Relative Changes to Baseline in levels of IL-23 effector proteins in biopsy tissue will be measured.

CONTACTS AND LOCATIONS:
Overall Officials: Janssen Research & Development, LLC Clinical Trial, Study Director — Janssen Research & Development, LLC
Locations (32):
- United States (18):
  - Mayo Clinic, Phoenix, Arizona
  - City of Hope, Duarte, California
  - Yale University, New Haven, Connecticut
  - Mayo Clinic Jacksonville, Jacksonville, Florida
  - University of Miami, Miami, Florida
  - University of South Florida, Tampa, Florida
  - Ochsner Medical Center, New Orleans, Louisiana
  - Massachusetts General Hospital, Boston, Massachusetts
  - Dana Farber Cancer Institute, Boston, Massachusetts
  - Washington University School Of Medicine, St Louis, Missouri
  - Herbert Irving Comprehensive Cancer Center Columbia University Medical Center, New York, New York
  - Cleveland Clinic, Cleveland, Ohio
  - Wexner Medical Center at the Ohio State University, Columbus, Ohio
  - University of Pennsylvania - Perelman School of Medicine, Philadelphia, Pennsylvania
  - Fox Chase Cancer Center, Philadelphia, Pennsylvania
  - University of Texas MD Anderson Cancer Center, Houston, Texas
  - University of Utah Huntsman Cancer Institute, Salt Lake City, Utah
  - University of Washington, Seattle, Washington
- France (2):
  - Hopital Edouard Herriot - CHU Lyon, Lyon
  - APHM Hopital Timone, Marseille
- Germany (2):
  - Universitatsklinikum Bonn, Bonn
  - Universitatsklinikum Ulm, Ulm
- Sourasky MC, Tel Aviv, Israel
- Netherlands (3):
  - Academisch Medisch Centrum Universiteit van Amsterdam, Amsterdam
  - Leiden University Medical Center, Leiden
  - Erasmus MC, Rotterdam
- Poland (2):
  - Szpital Kliniczny im Heliodora Swiecickiego Uniwersytetu Medycznego im Karola Marcinkowskiego w Po, Poznan
  - Narodowy Instytut Onkologii im Marii Sklodowskiej Curie Panstwowy Instytut Badawczy, Warsaw
- Pan American Center for Oncology Trials LLC, Rio Piedras, Puerto Rico
- Spain (2):
  - Hosp Univ Vall D Hebron, Barcelona
  - Hosp Clinic de Barcelona, Barcelona
- Karolinska Universitetssjukhuset, Stockholm, Sweden

REFERENCES:
- [Derived] Stone JK, Mehta NA, Singh H, El-Matary W, Bernstein CN. Endoscopic and chemopreventive management of familial adenomatous polyposis syndrome. Fam Cancer. 2023 Oct;22(4):413-422. doi: 10.1007/s10689-023-00334-3. Epub 2023 Apr 29. PMID 37119510